CLINICAL TRIAL: NCT06931379
Title: Screening for Lactose Intolerance Among Patients With IBS Diarrhea Dominant
Brief Title: Screening of Lactose Intolerance Among IBS Patients Diarrhea Dominant
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Christina Shahat Ayoub, resident at the tropical medicine department, Assiut University
Other Study IDs: Screening of lactose intolera
Record Dates: First submitted 2025-04-09; First posted 2025-04-17 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Lactose Intolerance
Keywords: lactose intolerance; chronic diarrhea
MeSH Terms: conditions — Lactose Intolerance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult patients aged 18-70 years diagnosed as IBS diarrhea dominant: The target population comprises individuals who meet the following inclusion criteria:
  Adults aged between 18 and 70 years.
  Diagnosed with IBS diarrhea dominant
  Both males and females are eligible for participation.

SUMMARY:
This cross-sectional study aims to determine the prevalence of lactose intolerance among patients with chronic diarrhea, assess its correlation with age and gender, and evaluate common symptoms in affected patients. The study will collect demographic data, conduct lactose intolerance testing via PCR, and use a symptom questionnaire.

DETAILED DESCRIPTION:
The study is designed as a cross-sectional analysis conducted at a single healthcare center. Its primary objectives are:

To determine the point prevalence of lactose intolerance in patients suffering from chronic diarrhea (lasting more than four weeks).

To explore potential correlations between lactose intolerance and demographic factors such as age and gender.

To identify the most common symptoms associated with lactose intolerance in this patient population.

Methodology:

Data Collection: Demographic information (age, sex, medical history, and diarrhea duration) will be gathered.

Lactose Intolerance Testing: Polymerase Chain Reaction (PCR) will be employed to diagnose lactose intolerance.

Symptom Questionnaire: A standardized questionnaire will be administered to document symptoms like abdominal pain, bloating, flatulence, diarrhea, and nausea.

ELIGIBILITY:
Inclusion Criteria:

* All Patients with IBS diarrhea dominant type meet Rome criteria attending at Al-Rajhy University Hospital during 6 months (from march to September). A patient must have recurrent abdominal pain (at least 1 day per week in the last 3 months) associated with at least two of the following:

  1. Related to defecation (pain improves or worsens with bowel movements).
  2. Change in stool frequency (diarrhea or constipation).
  3. Change in stool form (appearance) (loose, watery, hard, or lumpy).
* Patients aged >18 years.
* Both males and females

Exclusion Criteria:

* -patient aged<18 years old.
* Patients with chronic diarrhea don't meet Rome criteria
* patients with malignancies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18-70 years diagnosed with chronic diarrhea lasting more than four weeks. Both male and female participants are included. Participants will be recruited from a single healthcare center. They will undergo comprehensive assessments, including demographic profiling, medical history review, and diagnostic testing for lactose intolerance using PCR. The diversity in age and gender ensures that potential correlations with these variables can be analyzed.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Prevalence data on lactose intolerance in patients with IBS diarrhea dominant. | 1 year
  The primary outcome is to determine the percentage of patients with chronic diarrhea who test positive for lactose intolerance using PCR testing.